CLINICAL TRIAL: NCT03551535
Title: A Randomized Controlled Trial of the Feasibility and Adherence of a Prescribed, Monitored Home Exercise Program in High Risk Pregnant Women
Brief Title: Monitored Home Exercise in Pregnancy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study IRB approval expired
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00173362
Record Dates: First submitted 2018-05-03; First posted 2018-06-11 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2019-11

CONDITIONS: Exercise; Mobile Health; Pregnancy; Gestational Diabetes
Keywords: Wearable technology; Pregnancy; Exercise; Mobile Health
MeSH Terms: conditions — Motor Activity; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Experimental): Patients will be allocated to a physical activity intervention to be performed 3-5 days per week
  Interventions: Behavioral: Monitored, At-Home Exercise Intervention
- Control (No Intervention): Patients will receive standard counseling regarding activity recommendations in pregnancy

INTERVENTIONS:
Behavioral: Monitored, At-Home Exercise Intervention — Patients will be enrolled in the BurnAlong program as well as receive FitBit heart rate + activity monitors to track adherence rates to the prescribed exercise regimen on BurnAlong, with subsequent motivational interventions triggered if compliance varies from prescription
  Arms: Physical Activity Intervention

SUMMARY:
The Study Investigators intend to study the adherence to and effect of a prescribed, monitored at-home exercise regimen in a pregnant population at risk for gestational diabetes, with a specific goal of understanding factors relating to adoption and performance of regular, sustained physical activity.

DETAILED DESCRIPTION:
The obesity epidemic has affected the reproductive age population with a resultant increase in Gestational Diabetes Mellitus (GDM). Two to 10% of pregnant women are now diagnosed with gestational diabetes, imposing significant increased risk of maternal and fetal/neonatal morbidity and mortality.

Diabetes and obesity can both be combated by participating in daily physical activity, and has been shown to be beneficial for women of all ages, including women that are pregnant. The health benefits of exercise in pregnancy have been extensively studied, demonstrating improved pregnancy outcomes [both maternal (decreased gestational weight gain, decreased rates of cesarean section, and reduced rates of pregnancy induced complications such as hypertension and pre-eclampsia) and neonatal (reduction in proportion of large for gestational age infants)] with no evidence of harm when not contraindicated. Research should now focus on determining the most feasible, constructive, and efficient methods to improve fitness in pregnant women.

Pregnancy provides an ideal opportunity to focus on physical health and fitness; however, physical activity recommendations are rarely met and physical activity consistently decreases in pregnancy. With the development of mobile, technology-based interventions, at-home fitness regimens are now more accessible, thus reducing logistical constraints and burdens posed by traditional physical activity interventions. Moreover, the sustainability of at-home fitness regimens may be more successful long-term/post-intervention due to ease of engagement and more personalized motivational tools. Finally, wearable technology provides real-time feedback of progress and compliance to the intervention team, allowing improved monitoring of goals and compliance. In this way, contemporaneous, mobile health technology can maximize patient care by providing a novel, efficient, low burden, and scalable method to pursue pregnancy fitness, the economic implications of which could be significant.

The objective of this study is to determine the adherence to and effect of a prescribed, monitored at-home exercise regimen in a pregnant population at risk for gestational diabetes, with a specific goal of understanding factors relating to adoption and performance of regular, sustained physical activity.

There will be two arms of the study: an intervention group that will be enrolled in the BurnAlong program as well as receive FitBit heart rate + activity monitors to track adherence rates to the prescribed exercise regimen on BurnAlong, with subsequent motivational interventions triggered if compliance varies from prescription, and a comparison group who will receive standard obstetric care, which will include counseling about diet and exercise utilizing American Congress of Obstetricians and Gynecologists (ACOG) guidelines and literature, as well as a FitBit heart rate + activity monitor to track activity levels via step count. The project team will not interact with the comparison group regarding the patient's activity levels during the study duration.

A sample size of 25 women for each arm of the study (50 women total) will be recruited. Basic demographic data will be obtained for all enrolled subjects, including age, parity, pre-pregnancy BMI, family history of diabetes, history of GDM (and number of previously affected pregnancies), preterm birth history, and baseline activity level (type of job, exercise, hours of standing). All participants will be asked to fill out a physical activity in pregnancy readiness survey as well as a baseline, previously validated international physical activity questionnaire, which will be utilized for comparison to activity level data collected during the study period. All enrolled patients will receive a FitBit heart rate + activity monitor, which will provide overall activity data in the form of steps per day through the duration of the trial. Those randomized to the intervention group will also utilize the FitBit during exercise sessions to provide data on duration, heart rate, and intensity, all of which will confirm that exercise is being accomplished as prescribed. This immediate exercise compliance feedback will enable automated motivational factors to engage the patient and optimize their continued exercise participation. Data regarding mode of delivery as well as infant details will be collected by chart review by the research team. Long term follow up may be obtained via email surveys, thus patient emails will be obtained at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Singleton gestation
* History of gestational diabetes
* OR
* BMI ≥30
* OR
* Significant family history of diabetes (two or more first degree relatives with DM)

Exclusion Criteria:

* Non-English or non-Spanish speaking patients
* Women unwilling to provide consent
* Patients with current diagnosis of diabetes
* Multiple gestation
* Medical or pregnancy complications and/or comorbidities that preclude exercise in pregnancy
* Unwillingness to commit to the prescribed exercise program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant female participants only
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Adherence rate | 20 weeks
  Total number of performed exercise sessions divided by prescribed exercise sessions (3 per week at minimum)

SECONDARY OUTCOMES:
Gestational Diabetes | 20 weeks
  Development of Gestational diabetes as determined by routine 1 hour and then subsequent 3 hour glucose testing results
Maternal Weight Gain | 20 weeks
  measured in kilograms
Gestational age at delivery | One year
  Infant's gestational age at delivery
Rate of Cesarean delivery | One year
  measured as the number of cesarean deliveries per total number of deliveries
Infant weight | One year
  Infant weight in grams measured post delivery
Neonatal Apgar scores | 1, 5, and 10 minutes of neonatal life
  An assessment of neonatal wellbeing measured at 1, 5, and 10 minutes post-delivery, and is measured on a scale of 0-9, with 9 being the highest, and 0 being the lowest.
Neonatal Intensive Care Unit (NICU) Admission Rate | One year
  Rate of admission of infants post-delivery to the NICU
Neonatal hypoglycemia rates | One year
  Number of infants with hypoglycemia divided by the total number of delivered infants

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Sheffield, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Center for Chronic Disease Prevention and Health Promotion. National Diabetes Statistics Report, 2017.
- [Background] Impact of physical activity during pregnancy and postpartum on chronic disease risk. Med Sci Sports Exerc. 2006 May;38(5):989-1006. doi: 10.1249/01.mss.0000218147.51025.8a. PMID 16672855
- [Background] Borodulin KM, Evenson KR, Wen F, Herring AH, Benson AM. Physical activity patterns during pregnancy. Med Sci Sports Exerc. 2008 Nov;40(11):1901-8. doi: 10.1249/MSS.0b013e31817f1957. PMID 18845974
- [Background] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Background] World Health Organization. Global recommendations on physical activity for health. WHO (2010). Available at: http://www.who.int/dietphysicalactivity/publications/9789241599979/en. (Accessed: 23rd March 2018)
- [Background] Oguma Y, Shinoda-Tagawa T. Physical activity decreases cardiovascular disease risk in women: review and meta-analysis. Am J Prev Med. 2004 Jun;26(5):407-18. doi: 10.1016/j.amepre.2004.02.007. PMID 15165657
- [Background] ACOG Committee Opinion No. 650: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstet Gynecol. 2015 Dec;126(6):e135-e142. doi: 10.1097/AOG.0000000000001214. PMID 26595585
- [Background] Dempsey JC, Sorensen TK, Williams MA, Lee IM, Miller RS, Dashow EE, Luthy DA. Prospective study of gestational diabetes mellitus risk in relation to maternal recreational physical activity before and during pregnancy. Am J Epidemiol. 2004 Apr 1;159(7):663-70. doi: 10.1093/aje/kwh091. PMID 15033644
- [Background] Wang C, Wei Y, Zhang X, Zhang Y, Xu Q, Sun Y, Su S, Zhang L, Liu C, Feng Y, Shou C, Guelfi KJ, Newnham JP, Yang H. A randomized clinical trial of exercise during pregnancy to prevent gestational diabetes mellitus and improve pregnancy outcome in overweight and obese pregnant women. Am J Obstet Gynecol. 2017 Apr;216(4):340-351. doi: 10.1016/j.ajog.2017.01.037. Epub 2017 Feb 1. PMID 28161306
- [Background] Song C, Li J, Leng J, Ma RC, Yang X. Lifestyle intervention can reduce the risk of gestational diabetes: a meta-analysis of randomized controlled trials. Obes Rev. 2016 Oct;17(10):960-9. doi: 10.1111/obr.12442. Epub 2016 Jul 15. PMID 27417680
- [Background] Phelan S. Pregnancy: a "teachable moment" for weight control and obesity prevention. Am J Obstet Gynecol. 2010 Feb;202(2):135.e1-8. doi: 10.1016/j.ajog.2009.06.008. Epub 2009 Aug 15. PMID 19683692
- [Background] Evenson KR, Savitz DA, Huston SL. Leisure-time physical activity among pregnant women in the US. Paediatr Perinat Epidemiol. 2004 Nov;18(6):400-7. doi: 10.1111/j.1365-3016.2004.00595.x. PMID 15535815
- [Background] Gaston A, Cramp A. Exercise during pregnancy: a review of patterns and determinants. J Sci Med Sport. 2011 Jul;14(4):299-305. doi: 10.1016/j.jsams.2011.02.006. Epub 2011 Mar 21. PMID 21420359
- [Background] Ning Y, Williams MA, Dempsey JC, Sorensen TK, Frederick IO, Luthy DA. Correlates of recreational physical activity in early pregnancy. J Matern Fetal Neonatal Med. 2003 Jun;13(6):385-93. doi: 10.1080/jmf.13.6.385.393. PMID 12962263
- [Background] Poudevigne MS, O'Connor PJ. A review of physical activity patterns in pregnant women and their relationship to psychological health. Sports Med. 2006;36(1):19-38. doi: 10.2165/00007256-200636010-00003. PMID 16445309
- [Background] Oostdam N, van Poppel MN, Wouters MG, Eekhoff EM, Bekedam DJ, Kuchenbecker WK, Quartero HW, Heres MH, van Mechelen W. No effect of the FitFor2 exercise programme on blood glucose, insulin sensitivity, and birthweight in pregnant women who were overweight and at risk for gestational diabetes: results of a randomised controlled trial. BJOG. 2012 Aug;119(9):1098-107. doi: 10.1111/j.1471-0528.2012.03366.x. Epub 2012 May 23. PMID 22616913
- [Background] Olander EK, Atkinson L. Obese women's reasons for not attending a weight management service during pregnancy. Acta Obstet Gynecol Scand. 2013 Oct;92(10):1227-30. doi: 10.1111/aogs.12195. Epub 2013 Jul 5. PMID 23763541
- [Background] Sui Z, Turnbull DA, Dodd JM. Overweight and obese women's perceptions about making healthy change during pregnancy: a mixed method study. Matern Child Health J. 2013 Dec;17(10):1879-87. doi: 10.1007/s10995-012-1211-8. PMID 23263891
- [Background] Lau Y, Klainin-Yobas P, Htun TP, Wong SN, Tan KL, Ho-Lim ST, Chi C, Tsai C, Ong KW, Shorey S, Tam WSW. Electronic-based lifestyle interventions in overweight or obese perinatal women: a systematic review and meta-analysis. Obes Rev. 2017 Sep;18(9):1071-1087. doi: 10.1111/obr.12557. Epub 2017 May 22. PMID 28544551